CLINICAL TRIAL: NCT04165538
Title: Safety and Effectiveness of Clopidogrel Withdrawal Time Guided by Thromboelastography in Elderly Patients With Hip Fracture
Brief Title: Thromboelastography (TEG) and Clopidogrel Withdrawal Time in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-324
Record Dates: First submitted 2019-10-16; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Hip Fracture
Keywords: Hip Fracture; Clopidogrel; Withdrawal; surgical timing; Thromboelastogram
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEG group (Experimental)
  Interventions: Procedure: Thrombelastograph and surgical timing
- Non-TEG group (No Intervention)

INTERVENTIONS:
Procedure: Thrombelastograph and surgical timing — Patients in the TEG group will undergo a Thrombelastograph test after admission, and the timing of operation will be determined according to the results of the test, that is, 1 day, 3 days and 5 days later respectively for patients with ADP-induced platelet-fibrin clot strength (MAADP) of > 50 mm, 30-50 mm and < 30 mm. For Non-TEG patients, the drug withdrawal time is determined by the doctor in charge according to the clinical routine, generally about one week.
  Arms: TEG group

SUMMARY:
In the elderly patients with hip fracture, some often take antiplatelet drugs such as clopidogrel due to the ischemic cardiovascular or cerebrovascular diseases. In traditional practice, these patients often need to stop medication for 5-7 days before surgery. But on the other hand, delayed surgery will lead to a significant increase in fracture related complications. Therefore, the appropriate time for drug withdrawal is particularly important in this population.

Thromboelastography is a monitoring method that can accurately judge the anticoagulation status of patients. We hope to use thromboelastography to guide the time of drug withdrawal, shorten the time of drug withdrawal as much as possible, and reduce the incidence of fracture related complications without increasing the risk of massive hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture and operation
* taking clopidogrel for more than one week before injury, with or without taking aspirin at the same time

Exclusion Criteria:

* high energy injury (such as traffic accident, falling from height), bilateral hip fracture, multiple fractures or injuries, pathological fracture
* malignant tumor patients
* hormone users
* patients with recent active bleeding or bleeding ulcer
* primary or secondary coagulation dysfunction or depression caused by other reasons than taking antiplatelet drugs (for example, taking warfarin)
* patients with other acute or unstable diseases requiring delayed surgery (acute heart failure, myocardial infarction, cerebral infarction, cerebral hemorrhage, severe pulmonary infection, deep vein thrombosis or pulmonary embolism, etc.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Estimated red blood cell loss | From admission when the first blood routine will be obtained to discharge when the last blood routine will be obtained, up to postoperative day 7.
  The amount of red blood cell loss estimated by blood routine changes

SECONDARY OUTCOMES:
Blood transfusion | From admission when the first blood routine will be obtained to discharge when the last blood routine will be obtained, up to postoperative day 7.
  Red blood cell infusion volume

OTHER OUTCOMES:
Length of stay | from admission to discharge,up to one year after operation
  Total length of stay
Mortality | within one year after operation
  One year all-cause mortality
Cerebrovascular accident | within one year after operation
  Ischemic brain disease
Acute coronary syndrome | within one year after operation
  Ischemic heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Director — Zhejiang University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR